CLINICAL TRIAL: NCT06910826
Title: Explaining Spinal Anesthesia to Pregnant Women: A Visual Approach to Overcoming Fears
Brief Title: Visual Education for Spinal Anesthesia Acceptance
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. Prof, Istinye University
Other Study IDs: haseki broşür
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Incidence of Spinal Anesthesia Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Primary outcome: To determine the incidence of spinal anesthesia preference after exposure to the visual information catalog.

Secondary outcomes: To analyze independent (age, education, profession, previous experiences) and dependent (fear, anxiety) factors influencing patient choices.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45
* who are undergoing elective cesarean sections
* and classified as ASA I-II according to the American Society of Anesthesiologists (ASA) scale

Exclusion Criteria:

* patients under 18 or over 45 years old,
* emergency cesareans,
* preeclampsia,
* cardiovascular disorders,
* fetal abnormalities,
* those not receiving spinal anesthesia or converted to general anesthesia during surgery,
* those who refuse to participate in the study,
* hospital clinical or administrative staff,
* patients with psychiatric disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Study Population: The study will include 318 pregnant women aged 18-45 who are undergoing elective cesarean sections and classified as ASA I-II according to the American Society of Anesthesiologists (ASA) scale.
Sampling Method: Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
incidence of spinal anesthesia preference | 4 MONTH
  To determine the incidence of spinal anesthesia preference after exposure to the visual information catalog

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emadi SA, Gholipour Baradari A, Khademloo M, Abotorabi M, Hassanzadeh Kiabi F. Evaluating patients' choice of general and spinal anesthesia for elective cesarean section and associated factors: a descriptive study. Ann Med Surg (Lond). 2023 Jan 12;85(1):6-12. doi: 10.1097/MS9.0000000000000010. eCollection 2023 Jan. PMID 36742112
- [Background] Shahid N, Rashid AM. Knowledge, fear and acceptance rate of spinal anesthesia among pregnant women scheduled for cesarean section: a cross-sectional study from a tertiary care hospital in Karachi. BMC Anesthesiol. 2024 Nov 12;24(1):408. doi: 10.1186/s12871-024-02736-x. PMID 39533188